CLINICAL TRIAL: NCT00672152
Title: A Phase I Study of WT1 Peptides to Induce Anti-Leukemia Immune Responses Following Autologous or Allogeneic Transplantation for AML, CmML, ALL, MDS, and B Cell Malignancies
Brief Title: A Phase I Study of WT1 Peptides to Induce Anti-Leukemia Immune Responses Following Transplantation
Acronym: WT-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Michael Morse, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Morse, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001360
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Acute Myelogenous Leukemia (AML); Chronic Myelogenous Leukemia (CML); Acute Lymphoblastic Leukemia (ALL); Myelodysplastic Syndrome (MDS); B Cell Malignancies
Keywords: Autologous transplantation; Allogeneic transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A-WT1 derived peptides (Experimental): Wilms' tumor gene 1 (WT1) derived peptides consisting of 0.3mg (cohort 1) or 1mg (cohort 2) of each of the following peptides mixed with 1ml Montanide ISA 51 and 100mcg Granulocyte-macrophage colony-stimulating factor (GM-CSF) in a total volume of 2ml:
  * WT peptide #1: (human leukocyte antigen) HLA-A2 restricted: RMFPNAPYL
  * WT peptide #2: HLA-A24 restricted: CMTWNQMNL
  * WT peptide #3: HLA-DR15 restricted: QARMFPNAPYLPSCL
  * WT peptide #4: HLA-DRw53 restricted: LKGVAAGSSSSVKWT
  Immunization with the peptide pools will be given as 200 microliter intradermal and 1.8ml subcutaneously in opposite thighs.
  Interventions: Biological: WT1 derived peptides

INTERVENTIONS:
Biological: WT1 derived peptides — WT1 derived peptides consisting of 0.3mg (cohort 1) or 1mg (cohort 2) of each of the following peptides mixed with 1ml Montanide ISA 51 and 100mcg GM-CSF in a total volume of 2ml:
  * WT peptide #1: HLA-A2 restricted: RMFPNAPYL
  * WT peptide #2: HLA-A24 restricted: CMTWNQMNL
  * WT peptide #3: HLA-DR15 restricted: QARMFPNAPYLPSCL
  * WT peptide #4: HLA-DRw53 restricted: LKGVAAGSSSSVKWT
  Immunization with the peptide pools will be given as 200 microliter intradermal and 1.8ml subcutaneously in opposite thighs.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of administering Wilms tumor gene 1 (WT1) cancer peptides. Cancer peptides are short pieces of protein that are made in a laboratory to be like the peptides that can be found in cancer. These peptides are intended to be given as a "vaccine" to activate the immune cells in a person to attack his/her cancer. These peptides are mixed with an oily substance called Montanide ISA-51 and a white cell growth factor called Granulocyte-macrophage colony-stimulating factor (GM-CSF) which may help make the immune response stronger.

DETAILED DESCRIPTION:
Two subgroups with 2 dose cohorts of up to 6 patients each will be enrolled in this exploratory study in order to attempt to obtain immunologic and clinical data on patients with a variety of hematologic malignancies and amongst those in remission and early relapse. The 2 subgroups of patients will be treated with different schemas depending upon whether they are undergoing or have undergone autologous or allogeneic stem cell transplantation.

For the autologous transplant patients: Immune monitoring will require 90ml peripheral blood before the first immunization, 3-5 ml from the leukapheresis product, 40-90ml peripheral blood before the 4th immunization immunizations, after the last immunization (week 6-8), and at the discretion of the immune monitoring lab, every two months if immunizations are continued.

For the allogeneic transplant patients: Immune monitoring will require 90ml peripheral blood before the first immunization, 40-90ml peripheral blood before the 4th immunization immunizations, after the last immunization (week 6-8), and at the discretion of the immune monitoring lab, every two months if immunizations are continued.

Subjects will be monitored with blood pressure, temperature, and pulse, pre-injection, at 15 and 30 minutes after injection, prior to being allowed to leave the clinic. Diphenhydramine 50 mg, solumedrol 100 mg, and epinephrine 1:1000 (1 mL) must be available bedside (or a clinic code cart must be available). If hypotension (SBP <90mmHg for patients with baseline SBP > 110mmHg or > 20 mmHg decrease for those with baseline SBP< 110 mmHg), urticaria or orofacial or laryngeal edema or bronchospasm occurs, an IV line will be placed and the diphenhydramine 50 mg, solumedrol 100 mg, and epinephrine 1:1000 sq are recommended. In this event, patients will be transported emergently to the emergency room if stabilized or the code team will be contacted if patients continue to have progression of symptoms or worsening hypotension. For fever>101.5, acetaminophen 650 mg may be given orally.

ELIGIBILITY:
Inclusion Criteria:

There are two subgroups of patients: Those undergoing autologous stem cell transplantation and those undergoing allogeneic stem cell transplantation.

Autologous transplant subgroup:

-Patients with the following hematologic malignancies (AML, CML, ALL, B cell malignancies, and myelodysplastic syndrome) who will be undergoing autologous stem cell transplantation.

Allogeneic transplantation subgroup:

-Patients with the following hematologic malignancies (AML, CML, ALL, B cell malignancies, and myelodysplastic syndrome) who have undergone allogeneic stem cell transplantation. There is no limitation on whether myeloablative or non-myeloablative chemotherapy is administered. A 3/6 or greater match is required for patients who have had an allogeneic stem cell transplant.

Both subgroups:

* Subject must be one of the following HLA types: HLA A2, A24, DR15 or DRw53 (includes HLA-DR4, -DR7, and DRw9)
* Karnofsky performance status must be greater than or equal to 70%.
* Age ≥ 18 years.
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
* Patient must agree to use adequate contraception defined as: for women, one of the following (1) surgical sterilization, (2) approved hormonal contraceptives (such as birth control pills, Depo-Provera, or Lupron Depot), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD); for men, one of the following: (1) surgical sterilization, or (2) a condom used with a spermicide.
* In order to receive their immunizations, subjects should be:

For autologous transplants:

* At least 2 weeks from prior chemotherapy.
* Injections 1 and 2 must be completed prior to administration of any growth factor mobilization
* Injections 3, 4, 5, and 6, to resume 2 or more weeks from the time of their stem cell infusion if there has been no Grade 3 or 4 non-hematologic, major organ toxicity within the preceding 1 week. Non-major organ toxicities must have resolved to grade 2 or less.

For allogeneic transplants,

* At least 2 weeks from the time of their stem cell infusion.
* Without Grade 3 or 4 non-hematologic major organ toxicity within the preceding 1 week; non major organ toxicities must have resolved to grade 2 or less.
* We will require demonstration of >50% donor myeloid hematopoiesis, based on microsatellite polymorphisms, prior to enrolling the patients with MDS on the study.

  * Adequate laboratory data as follows:

Hematologic function: WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (may transfuse or use erythropoietin to achieve this level), platelets ≥ 50,000/microliter ((may transfuse).

Renal and hepatic function: serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except a bilirubin of <2.0 will be permitted for patents with Gilbert's syndrome), SGOT/SGPT < 2 x upper limit of normal.

* Subjects must have a CD4+ count is > 200/mm. There is no specified requirement for CD8+ T cell count.
* Urine protein/creatinine ratio (UPC) must be less than 1.

Exclusion Criteria:

* Corticosteroid (greater than 10mg per day of prednisone or an equipotent dose of another corticosteroid) or other immunosuppressive therapy within the prior 1 week.
* Pregnant women and nursing mothers.
* Current or prior history of brain metastases.
* More than 12 months since their stem cell transplant.
* HIV +, hepatitis BsAg +, Hepatitis C Ab+.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility | 2 years
  To determine the safety and feasibility of administering WT1 peptides to subjects who have undergone autologous or allogeneic stem cell transplantation for AML, CML, ALL, B cell malignancies and myelodysplastic syndrome.

SECONDARY OUTCOMES:
Immune Response | 2 years
  To evaluate the immune response to immunizations.
Efficacy (PFS and OS) | 2 years
  To obtain preliminary data on efficacy (PFS and OS) following immunization in those with available data.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Morse, MD, Principal Investigator — Duke University; Amy Hobeika, PhD, Study Director — Duke University; Nelson Chao, MD, Principal Investigator — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States